CLINICAL TRIAL: NCT01085877
Title: An Open Randomized Two-Way Cross-Over Comparative Bioavailability Study to Compare the Extent of Systemic Absorption of Estradiol After a Single Dose Treatment With Two 25 mcg Estradiol Vaginal Tablet Formulations Administered in Postmenopausal Women With Vaginal Atrophy
Brief Title: Comparison of Two Vaginal Tablets, Produced at Different Sites, in Postmenopausal Women With Atrophic Vaginitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VAG-3821; U1111-1113-4908 (Other: WHO); 2009-017034-50 (EudraCT Number)
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Menopause; Postmenopausal Vaginal Atrophy
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trial part 1 (Active Comparator)
  Interventions: Drug: estradiol, 25 mcg
- Trial part 2 (Experimental)
  Interventions: Drug: estradiol, 25 mcg

INTERVENTIONS:
Drug: estradiol, 25 mcg — Single dose of vaginal tablet containing 25 mcg estradiol (Production site A) followed by another single dose of vaginal tablet containing 25 mcg estradiol (Production site B)
  Arms: Trial part 1
Drug: estradiol, 25 mcg — Single dose of vaginal tablet containing 25 mcg estradiol (Production site B) followed by another single dose of vaginal tablet containing 25 mcg estradiol (Production site A)
  Arms: Trial part 2

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the absorption of estradiol after a single dose of two 25 mcg estradiol vaginal tablets, produced at two different production sites, in postmenopausal women with atrophic vaginitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to use the German language, spoken and written
* Postmenopausal women: 5 years or more after last menstruation; or both ovaries surgically removed 2 years or more prior to trial start
* Availability of a normal mammogram within 1 year prior to trial start
* Good general health
* No significant illnesses that could interfere with the subject's participation in the trial, based on the judgment of the physician

Exclusion Criteria:

* Known or suspected allergy to estradiol or related products
* Known, suspected or past history of breast cancer
* Abnormal genital bleeding
* Previous oestrogen and/or progestin hormone replacement therapy
* Use of any type of vaginal or vulvar preparations, e.g. pessaries, contraceptive sponges, douches, vaginal moisturizers, or other non-oestrogenic medications including K-Y jelly etc., 1 month prior to first planned drug administration
* Hot flushes which require systemic hormone replacement treatment
* Known insulin dependent or non-insulin dependent diabetes mellitus
* Systolic blood pressure (BP) of more than 160 mm Hg and/or diastolic BP or more than 100 mm Hg, currently treated or untreated
* Active deep venous thrombosis or thromboembolic disorders or a history of these conditions
* Active arterial thrombosis or a documented history of this condition
* Known or suspected liver and/or kidney impairment based on medical history, physical examination, and/or laboratory results
* Known HIV infection based on laboratory result
* Porphyria
* Body Mass Index (BMI) above 30.0 kg/m2
* Cervical smear presenting PAP of more than class II
* Known or suspected vaginal infection requiring further treatment
* Known alcohol or drug abuse, heavy smoking (more than 20 cigarettes a day)
* Currently using steroid hormones (except topical or inhalation glucocorticoid preparations) and drugs known to significantly influence oestrogen metabolism such as barbiturates, phenytoin, rifampicin, carbamazepine
* Subject who has participated in any other trial involving other investigational products within the last 30 days prior to the first planned drug administration

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC(0-t)), maximal concentration (Cmax) of estradiol after baseline correction | from dosing to day 4

SECONDARY OUTCOMES:
Number of adverse events and local tolerability | from dosing to day 4

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Mainz, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com